CLINICAL TRIAL: NCT00916396
Title: Dehydroepiandrosterone (DHEA) Treatment in Women and Men Experiencing Hypoactive Sexual Desire Disorder: Modulation of Sexual Libido by Androgens and Neurosteroids
Brief Title: Dehydroepiandrosterone (DHEA) Treatment in Women and Men Experiencing Hypoactive Sexual Desire Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Dr. Miki Bloch, Tel Aviv medical center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: tasmc-09-MB-158-ctil
Record Dates: First submitted 2009-06-07; First posted 2009-06-09 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2009-11

CONDITIONS: Hypoactive Sexual Desire Disorder
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- real drug (Active Comparator)
  Interventions: Drug: Dehydroepiandrosterone
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Dehydroepiandrosterone — 100 mg of DHEA a day (50 mg twice a day) for six weeks
  Other Names: DHEA
  Arms: real drug
Drug: placebo — 100 mg of Placebo a day (50 mg twice a day) for six weeks
  Arms: placebo

SUMMARY:
Hypoactive Sexual Desire Disorder (HSDD) is a common syndrome characterized by low sexual desire causing marked distress. The involvement of DHEA in sexual function is unknown, however, DHEA treatment increased desire in depressed subjects. In the current research, we will treat 45 women and men suffering from low sexual desire with DHEA or placebo for 6 weeks. The study's primary goal is to determine the effect of DHEA treatment on sexual desire, and to find if there is a connection between levels of hormones and change in desire. Outcome measures will include hormonal levels and psychological state. Our secondary goal is to compare baseline hormones measures in individuals with low sexual desire to normal controls. For that purpose we will measure the hormonal baseline levels among 20 normal subjects.

DETAILED DESCRIPTION:
Hypoactive Sexual Desire Disorder (HSDD) is a very common syndrome in adult women and men, characterized by a severe deficiency in the desire for sexual activity, causing marked distress. There is some data that androgens such as testosterone have some beneficial effect in this condition. DHEA is a neurosteroid that is metabolized into testosterone and estrogen, both of assumed importance in the regulation of sexual libido. The direct involvement of DHEA in the regulation of sexual function is unknown, however, DHEA treatment improved libido in midlife-onset depressed subjects. In this study, we will treat women and men suffering from HSDD with DHEA. The study's first objective is to determine the effect of DHEA treatment on sexual libido in menopausal women and both young and mid-aged men. The secondary objective is to compare baseline measures of DHEA, androgens, and other neurosteroids, in individuals with HSDD to controls. Furthermore, we will investigate possible correlations between plasma and urine levels of several neurosteroids and change in measures of libido. Fifty women and men diagnosed with HSDD will be treated with either 100 mg of DHEA or placebo for 6 weeks, in a double-blind, placebo-controlled study. Outcome measures will include several 17-Ketosteroids, DHEAS and bioavailable testosterone. Psychological outcome measures will include sexual function, mood and well-being. Twenty controls without HSDD will also be recruited to determine and compare their baseline levels of neurosteroids.

ELIGIBILITY:
Inclusion Criteria:

* Woman participating in the research will be in the menopausal phase or after it (above a year in postmenopause)aged 65 and below. Man age range will be 18 - 65.

Exclusion Criteria:

* Individuals suffering from a significant systemic illness, hormonal illness, alcoholism, drug abuse, major depression, "Mano/matroagia" or hypogonadism. Additionally, individuals treated with androgens, antidepressant or any other medication which may cause a disorder in sexual desire.
* Man diagnosed as suffering from prostate carcinoma, BHP or will show PSA levels above 2.5 will not be included.
* Woman treated with HRT or suffering from any of the following diseases will not be included: breast carcinoma, ovarian or uterus cancer or with a first grade family history of one of the mentioned.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-06; Primary Completion 2011-01 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
blood and urine tests | beginning of treatment, and after six weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Miki Bloch, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Aviv Medical Center, Tel Aviv, Israel

REFERENCES:
- [Derived] Bloch M, Meiboom H, Zaig I, Schreiber S, Abramov L. The use of dehydroepiandrosterone in the treatment of hypoactive sexual desire disorder: a report of gender differences. Eur Neuropsychopharmacol. 2013 Aug;23(8):910-8. doi: 10.1016/j.euroneuro.2012.09.004. Epub 2012 Oct 18. PMID 23084789